CLINICAL TRIAL: NCT07035704
Title: De-Risking Metabolic, Environmental and Behavioral Determinants of Obesity in Children, Adolescents and Young Adults
Brief Title: Prevent and Reverse Obesity in Children, Adolescents and Young Adults
Acronym: PasGras
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: piero portincasa (Other)
Collaborators: University of Bari Aldo Moro (Other); Uppsala University (Other); Fundació Eurecat (Other); ADPD (Unknown); University of Coimbra (Other); AGDCENTRO ASSOCIACAO DE GINASTICA DO CENTRO (Unknown); INSTITUTO POLITECNICO DE VIANA DE CASTELO (Unknown); Consiglio Nazionale delle Ricerche, Italy (Unknown); Technical University of Munich (Other); MEDIAGNOST GESELLSCHAFT FUR FORSCHUNG UND HERSTELLUNG VON DIAGNOSTIKA GMBH (Unknown); Martin-Luther-Universität Halle-Wittenberg (Other); THE EUROPEAN SOCIETY FOR CLINICAL INVESTIGATION (Unknown); INSTYTUT BIOLOGII DOSWIADCZALNEJ IM. M. NENCKIEGO POLSKIEJ AKADEMII NAUK (Unknown); King's College London (Other)
Responsible Party: Sponsor-Investigator, piero portincasa, Professor, University of Bari
Organization: University of Bari (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PasGras 2025
Record Dates: First submitted 2025-06-10; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-12

CONDITIONS: Overweight (BMI > 25)
Keywords: MeD diet, Healthy life, obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: This will be a 12-month, controlled, randomized, multicenter clinical study with five arms.
  The suggested study design will allow to compare different outcomes in subjects included in each treatment arm.
  The study will involve a total of 250 participants from four different centers in four European countries (Spain, Italy, Sweden, and Portugal). The subjects will be assessed at baseline and monitored for 12 months follow-up. Enrolled subjects will be randomly assigned to one of the following three treatment groups.
  * Group 1: MeD personalized plan: will receive counselling and personalized dietary strategy aimed at increasing the adherence to Mediterranean diet by means of use of visual communication (e.g., comics, cartoons, videos) and digital tools (i.e., games, apps), including a physical activity program with a personal trainer.
  * Group 2: MeD enriched with mushrooms or other dietary supplements: will receive the MeD personalized plan plus commercial mushrooms or other suppleme
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MeD personalized plan (Active Comparator): Patients will receive counselling and personalized dietary strategy aimed at increasing the adherence to Mediterranean diet by means of use of visual communication (e.g., comics, cartoons, videos) and digital tools (i.e., games, apps), including a physical activity program with a personal trainer
  Interventions: Dietary Supplement: MeD enriched with mushrooms; Dietary Supplement: MeD enriched the Lebanese herbal mixture Za'atar
- MeD in combination with semaglutide (Active Comparator): Patients will receive counselling and personalized dietary strategy aimed at increasing the adherence to Mediterranean diet by means of use of visual communication (e.g., comics, cartoons, videos) and digital tools (i.e., games, apps), including a physical activity program with a personal trainer + semaglutinine or compatible treatment
  Interventions: Dietary Supplement: MeD Diet + semaglutinine or compatible treatment+ Za'atar or Mushroom (to be defined)

INTERVENTIONS:
Dietary Supplement: MeD enriched with mushrooms — Patients will receive the MeD personalized plan plus commercial mushrooms
  Arms: MeD personalized plan
Dietary Supplement: MeD enriched the Lebanese herbal mixture Za'atar — Patients will receive the MeD personalized plan plus natural products/extracts of endemic plants (olive oil, herbs like Lebanese Za'atar).
  Arms: MeD personalized plan
Dietary Supplement: MeD Diet + semaglutinine or compatible treatment+ Za'atar or Mushroom (to be defined) — Patients will receive counselling and personalized dietary strategy aimed at increasing the adherence to Mediterranean diet by means of use of visual communication (e.g., comics, cartoons, videos) and digital tools (i.e., games, apps), including a physical activity program with a personal trainer + semaglutinine or compatible treatment+ Za'atar or Mushroom (to be defined)
  Arms: MeD in combination with semaglutide

SUMMARY:
Obesity and overweight are non-communicable diseases with an increasing incidence in children, adolescents, and adults. International efforts to reverse the current epidemiological trend of rising overweight, obesity, and related diseases have so far been insufficient to achieve this goal. Therefore, a change in strategy-both at the individual and public health levels-is urgently needed.

Searching the litterature, there are currently no studies employing a comprehensive, personalized, and multi-level strategy to induce stable changes in dietary and lifestyle habits, while also conducting careful follow-up of outcomes and exploring the pathogenic mechanisms affecting metabolic pathways, pro-inflammatory and systemic conditions, and intestinal permeability in overweight and obese patients.

Evidence shows the beneficial effects of specific dietary patterns (e.g., the Mediterranean Diet) and a healthy lifestyle in reducing body/organ fat accumulation. However, a comprehensive evaluation of their effects-particularly following personalized strategies and careful follow-up-on the pathogenic mechanisms influencing cardiovascular and metabolic risk, pro-inflammatory status, and intestinal permeability in the medium-to-long term is still lacking.

DETAILED DESCRIPTION:
The study will enroll 200 adults overweight or obese patients (balanced by sex) attending the metabolic diseases outpatient clinic.

The MeD effects on the reduction of cardiometabolic risk in overweight and obese individuals originate beyond the nutritional component. The combination of personalized dietary and lifestyle treatments in the MeD setting can result in a greater strategy to reduce overweight, obesity and related cardiometabolic risk factors than the MeD alone.

Therefore, in the present study reaserchers hypothesize that the MeD associated with personalized dietary, lifestyle, and therapeutic strategies, including digital tools, a physical activity program, and under-explored MeD components such as mushrooms and the Lebanese herbal mixture "Za'atar", can increase the diet efficacy in tackling overweight and obesity.

Primary Objective: To identify and validate personalized interventions (tailored to individual risk) aimed at reducing health risks associated with overweight and obesity by targeting environmental, socio-cultural, and metabolic health determinants responsible for fat accumulation and related systemic diseases.

Secondary Objectives: To evaluate the nutritional and functional benefits of personalized dietary/lifestyle strategies on pathogenic factors influencing metabolic and pro-inflammatory status and intestinal permeability.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old overweight or obese men and women (BMI ≥ 25 kg/m2).
* Signed informed consent.
* Have a mobile phone, tablet, or computer with internet access.

Exclusion Criteria:

* Waist circumference > 150 cm
* Suffer from diabetes or other disorders of glucose metabolism
* Suffer from dyslipidemia or other alterations of lipid metabolism (LDL cholesterol ≥ 189 mg/dL and/or triglycerides ≥ 350 mg/dL).
* Present chronic gastrointestinal problems such as Crohn's disease or irritable bowel syndrome.
* Present any chronic or autoimmune disease in clinical manifestation such as hepatitis, hyper or hypothyroidism or metabolic diseases.
* Have a diagnosed liver disease other than steatotic liver disease.
* Taking supplements or multivitamin supplements or phototherapeutic products for weight loss that interfere with the study.
* Have taken antibiotics in the last 30 days.
* Follow a low-calorie diet and/or pharmacological treatment for weight loss.
* Being a smoker.
* Regular alcohol consumption (more than 4 Standard Drink Units (SDU) per day or 28 SDU per week.
* Have lost more than 3 kg of weight in the last 3 months.
* Suffering from eating disorders or psychiatric disorders.
* Present food intolerances and/or allergies related to the study products, such as allergy to edible mushrooms or fungal spores or to any of the components of the Lebanese herbal mixture Za'atar such as sesame seeds.
* Be pregnant or intend to become pregnant or be breastfeeding,
* Participate in or have participated in a clinical trial or nutritional intervention study in the last 30 days prior to inclusion in the study.
* No or limited access to the Internet.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Weight (Kg) | one year
  The primary outcome is weight loss

SECONDARY OUTCOMES:
Liver enzymes | one year
  Change in AST, ALT, and GGT
Fasting glucose | one year
  Change in glycemic profile
Lipid profile (TC, TG, LDL, HDL) | one year
  Change in Lipid profile
Abdominal fat storage | one year
  Change in abdominal fat depostion
Liver steatosis | one year
  Assessment of liver fat accumulation

OTHER OUTCOMES:
Inflammatory markers | One year
  Assessment of serum inflammatory markers such as Interleukins and cytokines
Gut Microbiota | one year
  Assessment of fecal gut microbiota composition

CONTACTS AND LOCATIONS:
Overall Officials: Piero Portincasa, PhD, Principal Investigator — University of Bari Aldo Moro
Locations (1):
- UniBa, Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No
Anonymised Data will be share ONLY among partners

REFERENCES:
- [Background] Portincasa P, Bonfrate L, Vacca M, De Angelis M, Farella I, Lanza E, Khalil M, Wang DQ, Sperandio M, Di Ciaula A. Gut Microbiota and Short Chain Fatty Acids: Implications in Glucose Homeostasis. Int J Mol Sci. 2022 Jan 20;23(3):1105. doi: 10.3390/ijms23031105. PMID 35163038
- [Background] Van Gorp H, Huang L, Saavedra P, Vuylsteke M, Asaoka T, Prencipe G, Insalaco A, Ogunjimi B, Jeyaratnam J, Cataldo I, Jacques P, Vermaelen K, Dullaers M, Joos R, Sabato V, Stella A, Frenkel J, De Benedetti F, Dehoorne J, Haerynck F, Calamita G, Portincasa P, Lamkanfi M. Blood-based test for diagnosis and functional subtyping of familial Mediterranean fever. Ann Rheum Dis. 2020 Jul;79(7):960-968. doi: 10.1136/annrheumdis-2019-216701. Epub 2020 Apr 20. PMID 32312770
- [Background] Rizzello CG, Portincasa P, Montemurro M, Di Palo DM, Lorusso MP, De Angelis M, Bonfrate L, Genot B, Gobbetti M. Sourdough Fermented Breads are More Digestible than Those Started with Baker's Yeast Alone: An In Vivo Challenge Dissecting Distinct Gastrointestinal Responses. Nutrients. 2019 Dec 4;11(12):2954. doi: 10.3390/nu11122954. PMID 31817104
- [Background] Cosola C, Rocchetti MT, di Bari I, Acquaviva PM, Maranzano V, Corciulo S, Di Ciaula A, Di Palo DM, La Forgia FM, Fontana S, De Angelis M, Portincasa P, Gesualdo L. An Innovative Synbiotic Formulation Decreases Free Serum Indoxyl Sulfate, Small Intestine Permeability and Ameliorates Gastrointestinal Symptoms in a Randomized Pilot Trial in Stage IIIb-IV CKD Patients. Toxins (Basel). 2021 May 5;13(5):334. doi: 10.3390/toxins13050334. PMID 34063068
- [Background] Molina-Molina E, Shanmugam H, Di Ciaula A, Grattagliano I, Di Palo DM, Palmieri VO, Portincasa P. (13C)-Methacetin breath test provides evidence of subclinical liver dysfunction linked to fat storage but not lifestyle. JHEP Rep. 2020 Nov 4;3(1):100203. doi: 10.1016/j.jhepr.2020.100203. eCollection 2021 Feb. PMID 33490935
- [Background] Di Ciaula A, Baj J, Garruti G, Celano G, De Angelis M, Wang HH, Di Palo DM, Bonfrate L, Wang DQ, Portincasa P. Liver Steatosis, Gut-Liver Axis, Microbiome and Environmental Factors. A Never-Ending Bidirectional Cross-Talk. J Clin Med. 2020 Aug 14;9(8):2648. doi: 10.3390/jcm9082648. PMID 32823983
- [Background] Vacca M, Celano G, Calabrese FM, Portincasa P, Gobbetti M, De Angelis M. The Controversial Role of Human Gut Lachnospiraceae. Microorganisms. 2020 Apr 15;8(4):573. doi: 10.3390/microorganisms8040573. PMID 32326636
- [Background] Bonfrate L, Di Palo DM, Celano G, Albert A, Vitellio P, De Angelis M, Gobbetti M, Portincasa P. Effects of Bifidobacterium longum BB536 and Lactobacillus rhamnosus HN001 in IBS patients. Eur J Clin Invest. 2020 Mar;50(3):e13201. doi: 10.1111/eci.13201. Epub 2020 Feb 12. PMID 31960952
- [Background] Di Palo DM, Garruti G, Di Ciaula A, Molina-Molina E, Shanmugam H, De Angelis M, Portincasa P. Increased Colonic Permeability and Lifestyles as Contributing Factors to Obesity and Liver Steatosis. Nutrients. 2020 Feb 21;12(2):564. doi: 10.3390/nu12020564. PMID 32098159
- [Background] Baldini F, Khalil M, Bartolozzi A, Vassalli M, Di Ciaula A, Portincasa P, Vergani L. Relationship between Liver Stiffness and Steatosis in Obesity Conditions: In Vivo and In Vitro Studies. Biomolecules. 2022 May 23;12(5):733. doi: 10.3390/biom12050733. PMID 35625660
- [Background] Faienza MF, Chiarito M, Molina-Molina E, Shanmugam H, Lammert F, Krawczyk M, D'Amato G, Portincasa P. Childhood obesity, cardiovascular and liver health: a growing epidemic with age. World J Pediatr. 2020 Oct;16(5):438-445. doi: 10.1007/s12519-020-00341-9. Epub 2020 Feb 4. PMID 32020441
- [Background] Di Ciaula A, Portincasa P. Diet and Contaminants: Driving the Rise to Obesity Epidemics? Curr Med Chem. 2019;26(19):3471-3482. doi: 10.2174/0929867324666170518095736. PMID 28521687
- [Background] Faienza MF, Wang DQ, Fruhbeck G, Garruti G, Portincasa P. The dangerous link between childhood and adulthood predictors of obesity and metabolic syndrome. Intern Emerg Med. 2016 Mar;11(2):175-82. doi: 10.1007/s11739-015-1382-6. Epub 2016 Jan 12. PMID 26758061
- [Background] Bonfrate L, Wang DQ, Garruti G, Portincasa P. Obesity and the risk and prognosis of gallstone disease and pancreatitis. Best Pract Res Clin Gastroenterol. 2014 Aug;28(4):623-35. doi: 10.1016/j.bpg.2014.07.013. Epub 2014 Jul 22. PMID 25194180
- [Background] Vecchie A, Dallegri F, Carbone F, Bonaventura A, Liberale L, Portincasa P, Fruhbeck G, Montecucco F. Obesity phenotypes and their paradoxical association with cardiovascular diseases. Eur J Intern Med. 2018 Feb;48:6-17. doi: 10.1016/j.ejim.2017.10.020. PMID 29100895
- [Background] Baldini F, Khalil M, Serale N, Voci A, Portincasa P, Vergani L. Extent and features of liver steatosis in vitro pave the way to endothelial dysfunction without physical cell-to-cell contact. Nutr Metab Cardiovasc Dis. 2021 Nov 29;31(12):3522-3532. doi: 10.1016/j.numecd.2021.08.032. Epub 2021 Aug 13. PMID 34629256
- [Background] Di Ciaula A, Bonfrate L, Krawczyk M, Fruhbeck G, Portincasa P. Synergistic and Detrimental Effects of Alcohol Intake on Progression of Liver Steatosis. Int J Mol Sci. 2022 Feb 27;23(5):2636. doi: 10.3390/ijms23052636. PMID 35269779
- [Background] Portincasa P, Bonfrate L, Khalil M, Angelis M, Calabrese FM, D'Amato M, Wang DQ, Di Ciaula A. Intestinal Barrier and Permeability in Health, Obesity and NAFLD. Biomedicines. 2021 Dec 31;10(1):83. doi: 10.3390/biomedicines10010083. PMID 35052763
- [Background] Yarnoz-Esquiroz P, Olazaran L, Aguas-Ayesa M, Perdomo CM, Garcia-Goni M, Silva C, Fernandez-Formoso JA, Escalada J, Montecucco F, Portincasa P, Fruhbeck G. 'Obesities': Position statement on a complex disease entity with multifaceted drivers. Eur J Clin Invest. 2022 Jul;52(7):e13811. doi: 10.1111/eci.13811. Epub 2022 May 12. PMID 35514242
- See also: PROJECT INFO AND DESCRIPTION — https://pasgras.eu/goals-and-impact